CLINICAL TRIAL: NCT04555694
Title: Intracanalicular Dexamethasone Used in Conjunction With Restasis (Cyclosporine Ophthalmic Emulsion) for the Treatment of Signs and Symptoms of Dry Eye Disease as Compared to Restasis With Lotemax (Loteprednol Etabonate Ophthalmic Suspension 0.5%) and Restasis Monotherapy.
Brief Title: Comparing Treatment of Dry Eye With Intracanalicular Dexamethasone, Restasis, and/or Lotemax
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Chester, OD (Other)
Responsible Party: Sponsor-Investigator, Thomas Chester, OD, Principal Investigator, Cleveland Eye Clinic
Organization: Cleveland Eye Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-2020-DexRes
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporine; Cyclosporins; Loteprednol Etabonate; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: 10 subjects will receive Restasis and Dextenza 10 subjects will receive Restasis and Lotemax 10 subjects will receive Restasis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Restasis and Lotemax (Active Comparator): 10 subjects will be receiving Restasis ophthalmic solution twice a day in both eyes and Lotemax ophthalmic solution twice a day in both eyes.
  Interventions: Drug: Cyclosporine; Drug: Loteprednol Etabonate
- Restasis and Dextenza (Active Comparator): 10 subjects will be receiving Restasis ophthalmic solution twice a day in both eyes, as well as receiving Dextenza insertion in both lower lids.
  Interventions: Drug: Cyclosporine; Drug: Dexamethasone Ophthalmic 0.4 Mg Ophthalmic Insert
- Restasis (Active Comparator): 10 subjects will be receiving Restasis ophthalmic solution twice a day in both eyes
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine — Used to increase tear production in patients who have dry eye caused by inflammation
  Other Names: Restasis
Drug: Loteprednol Etabonate — Used to treat inflammation of the eye
  Other Names: Lotemax
  Arms: Restasis and Lotemax
Drug: Dexamethasone Ophthalmic 0.4 Mg Ophthalmic Insert — Used to treat inflammation of the eye
  Other Names: Dextenza
  Arms: Restasis and Dextenza

SUMMARY:
This 6 month study seeks to compare the use of Intracanalicular Dexamethasone in conjunction with Restasis (cyclosporine ophthalmic emulsion) for the treatment of signs and symptoms of dry eye disease as compared to Restasis with Lotemax (loteprednol etabonate ophthalmic suspension 0.5%) and Restasis monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Signs and symptoms of Dry Eye Disease
* Consent to treat with topical immunomodulator
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Altered nasolacrimal flow of either acquired, induced, or congenital origin
* Hypersensitivity to dexamethasone
* Patients who have been on topical immunomodulating agents in the previous 3 months to their baseline visit
* Patient being treated with either topical, oral, or intravenous immunosuppressive agents, immunomodulating agents, or steroid (including NSAIDS)
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Eye Clinic, Brecksville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty patients were enrolled in the study. 10 patients in each treatment group.
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis
Started | 10; 20 Eyes | 10; 20 Eyes | 10; 20 Eyes
Completed | 10; 20 Eyes | 10; 20 Eyes | 10; 20 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Full Range); unit: years] | 59 [44 to 72] | 55 [32 to 78] | 62 [43 to 79] | 58 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 9 | 23
  Male | 2 | 4 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 10 | 8 | 7 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Ocular Surface Staining From Baseline
Description: The primary outcome measure was the mean corneal surface staining (guided by use of fluorescein and lissamine green) at weeks 4, 8 and 12 from baseline based on the National Eye Institute grading scale.
  Corneal fluorescein staining was scored from 0 to 3 on the scale (none, better to heavy, worse) in five regions of the cornea and summed for a total score of 0-15.
Time Frame: Baseline to Week 4, Week 8 and Week 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Eyes
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (Eyes) | 20 | 20 | 18
Score on a scale
  Baseline | 0.8 (1.5) | 0.6 (1.0) | 0.5 (0.5)
  Week 4 | 0.9 (0.9) | 0.6 (1.0) | 1.1 (1.4)
  Week 8 | 0.0 (0.0) | 0.5 (1.1) | 0.3 (0.6)
  Week 12 | 0.6 (1.0) | 0.7 (1.4) | 0.5 (0.7)

2. Secondary Outcome: Mean Conjunctival Staining
Description: The mean conjunctival staining (guided by use of lissamine green) at weeks 4, 8 and 12 from baseline based on the National Eye Institute grading scale.
  Conjunctival staining was scored from 0 to 3 on the scale (none, better to heavy, worse) in six regions of the cornea and summed for a total score of 0-18.
Time Frame: Baseline to Week 4, Week 8 and Week 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Eyes
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (Eyes) | 20 | 20 | 18
Score on a scale
  Baseline | 1.5 (1.8) | 0.5 (1.8) | 0.4 (0.6)
  Week 4 | 0.9 (1.4) | 0.3 (0.6) | 0.5 (0.7)
  Week 8 | 0.8 (1.8) | 0.4 (0.8) | 0.3 (0.6)
  Week 12 | 1.0 (1.6) | 0.8 (1.7) | 0.7 (1.4)

3. Secondary Outcome: Mean Schirmer Tear Test 1 Score
Description: Schirmer Tear Test 1 score, measuring tear production, as measured by a Schirmer's test strip with anesthetic (mm/5min on a strip 0-35mm. 0 mm is worse, >15 indicates normal production) at week 4, 8 and 12 from Baseline.
Time Frame: Baseline to Week 4, Week 8 and Week 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Eyes
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (Eyes) | 20 | 20 | 18
Score on a scale
  Baseline | 10.3 (7.2) | 14.9 (10.3) | 11.6 (10.5)
  Week 4 | 12.9 (9.1) | 15.4 (10.1) | 10.1 (8.5)
  Week 8 | 12.4 (8.4) | 15.8 (9.4) | 10.8 (6.4)
  Week 12 | 10.1 (6.0) | 12.3 (7.1) | 9.6 (5.5)

4. Secondary Outcome: Tear Breakup Time (Seconds)
Description: The time it takes (in seconds) for the tear film to break after blinking at Week 4, 8 and 12 from Baseline
Time Frame: Baseline to Week 4, Week 8 and Week 12
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Eyes
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (Eyes) | 20 | 20 | 18
Seconds
  Basline | 5.4 (1.5) | 6.6 (2.2) | 5.7 (3.3)
  Week 4 | 6.1 (2.8) | 8.0 (3.6) | 7.4 (3.7)
  Week 8 | 6.2 (2.2) | 7.7 (3.1) | 7.1 (3.4)
  Week 12 | 6.1 (2.4) | 7.7 (2.5) | 7.3 (3.6)

5. Secondary Outcome: Tear Osmolarity
Description: Tear osmolarity as measured by TearLab (275-307 is considered "homeostatic range") at Week 4, 8 and 12 from Baseline.
Time Frame: Baseline to Week 4, Week 8 and Week 12
Measure: Mean (Standard Deviation); unit: mOsM/L
Units Other Than Participants: Eyes
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (Eyes) | 20 | 20 | 18
mOsM/L
  Baseline | 311.3 (19.8) | 295.5 (17.4) | 306.9 (28.4)
  Week 4 | 307.7 (17.3) | 304.4 (30.1) | 307.9 (24.2)
  Week 8 | 300.1 (19.2) | 303.9 (22.1) | 295.3 (20.7)
  Week 12 | 304.4 (28.7) | 299.5 (16.2) | 304.6 (19.6)

6. Secondary Outcome: Meibomian Gland Scores
Description: Meibomian gland scoring on a scale of 1-4 (1 represents clear, liquid secretions and 4 is no secretions) in three regions (nasal, central, temporal) and summed for a single score between 3-12 at Week 4, 8 and 12 from baseline
Time Frame: Baseline to Week 4, Week 8 and Week 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Eyes
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (Eyes) | 20 | 20 | 18
Score on a scale
  Baseline | 7.1 (2.1) | 8.7 (2.4) | 9.2 (2.6)
  Week 4 | 6.7 (2.5) | 7.6 (1.8) | 7.2 (1.4)
  Week 8 | 6.3 (2.6) | 8.3 (2.0) | 8.2 (2.2)
  Week 12 | 6.0 (2.3) | 8.7 (2.0) | 7.3 (1.4)

7. Secondary Outcome: DEQ-5 Score
Description: Dry Eye Questionnaire-5 (5 questions about dry eye symptoms rated from 0, or never to 5, or constantly) total score of 0-22 with higher scores representing worse symptoms at weeks 4, 8 and 12 from baseline
Time Frame: Baseline to Week 4, Week 8 and Week 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: Eyes
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis
Number analyzed (Participants) | 10 | 10 | 9
Number analyzed (Eyes) | 20 | 20 | 18
Score on a scale
  Baseline | 14.4 (2.4) | 14.1 (4.0) | 14.4 (3.7)
  Week 4 | 11.0 (2.4) | 10.6 (4.6) | 12.2 (2.2)
  Week 8 | 9.1 (4.0) | 11.3 (4.5) | 10.6 (2.6)
  Week 12 | 10.2 (3.8) | 10.3 (6.3) | 9.4 (3.1)

ADVERSE EVENTS:
Time Frame: Baseline to Week 12
Arm/Group | Restasis and Lotemax | Restasis and Dextenza | Restasis
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 2/10 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Restasis and Lotemax (N=10) | Restasis and Dextenza (N=10) | Restasis (N=10)
2+ Injection at week 8 visit. (Eye disorders) | 0 | 1 | 0 — 2+ injection at week 8 visit. No treatment necessary. Improving upon exit.
Increased Corneal and Conjunctival Staining from Baseline (Eye disorders) | 0 | 1 | 0 — Increased corneal and conjunctival staining from baseline to exit visit. No treatment necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT04555694/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT04555694/SAP_001.pdf